CLINICAL TRIAL: NCT03378219
Title: Kevzara® (Sarilumab) Pregnancy Exposure Registry: An OTIS Pregnancy Surveillance Study
Brief Title: An Observational Study on Sarilumab-exposed Pregnancies
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS15155; U1111-1200-1947 (Registry Identifier: ICTRP)
Record Dates: First submitted 2017-12-15; First posted 2017-12-19 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis -Exposure During Pregnancy
MeSH Terms: interventions — sarilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Sarilumab-Exposed Cohort: Pregnant women exposed to Kevzara (sarilumab) for the treatment of an approved Kevzara (sarilumab) indication, for any number of days, at any dose, and at any time from the first day of the last menstrual period (LMP) up to and including the end of pregnancy
  Interventions: Drug: Sarilumab SAR153191 (REGN88)
- Cohort 2: Disease-matched Comparison Cohort: Pregnant women diagnosed with Kevzara (sarilumab) approved indication. Approximate frequency matched to the exposed group by disease indication, validated by medical records, who have not been exposed to Kevzara (sarilumab) any time in the current pregnancy, and have taken another biologic DMARD medication for their disease within 2 years before the current pregnancy and have an indication for such treatment at enrollment
- Cohort 3: Non-diseased Comparison Cohort: Healthy pregnant women not diagnosed with a Kevzara (sarilumab) indication and unexposed to Kevzara (sarilumab) during the course of the pregnancy

INTERVENTIONS:
Drug: Sarilumab SAR153191 (REGN88) — Pharmaceutical form:injection Route of administration: subcutaneous
  Other Names: Kevzara
  Groups: Cohort 1

SUMMARY:
Primary Objective:

To evaluate the relative risk of major structural birth defects, specifically a pattern of anomalies, in sarilumab-exposed pregnancies compared to disease-matched unexposed pregnancies.

Secondary Objective:

To evaluate the risk for sarilumab-exposure relative to the group of healthy pregnant women, and the effect of exposure on other adverse pregnancy and infants outcomes.

DETAILED DESCRIPTION:
Pregnant women enrolled in the study will participate for the duration of that pregnancy. Those who deliver at least one live born infant and the infants will participate for 1 year after delivery of that infant.

ELIGIBILITY:
Inclusion criteria:

* Cohort 1: Sarilumab-Exposed Cohort
* Currently pregnant, exposed to Kevzara (sarilumab) for approved indication
* Cohort 2: Disease-matched Comparison Cohort
* Currently pregnant, diagnosed with Kevzara (sarilumab) approved indication
* Cohort 3: Non-diseased Comparison Cohort
* Currently pregnant, not diagnosed with a Kevzara (sarilumab) indication and unexposed to Kevzara

Exclusion criteria:

First contact the Registry after prenatal diagnosis of any major structural defect or after pregnancy outcome is known (retrospective data).

Enrolled in this cohort study with a previous pregnancy. Cohort 1: Sarilumab-Exposed Cohort

* Exposed to Kevzara (sarilumab) for an indication other than a currently approved indication.
* Exposure to another biologic during pregnancy or within 10 weeks prior to the first day of LMP.
* Exposed to methotrexate, cyclophosphamide, chlorambucil, or mycophenolate mofetil in pregnancy (ie, at any time after the LMP), or leflunomide within two years prior to pregnancy unless a blood level for leflunomide below 0.02 mcg/mL has been documented prior to LMP before the pregnancy.
* Cohort 2: Disease-matched Comparison Cohort
* Exposure to any Kevzara (sarilumab) during pregnancy or within 10 weeks prior to the first day of the LMP.
* Exposed to methotrexate, cyclophosphamide, chlorambucil, or mycophenolate mofetil in pregnancy (ie, at any time after the LMP), or leflunomide within two years prior to pregnancy unless a blood level for leflunomide below 0.02 mcg/mL has been documented prior to LMP before the pregnancy.
* Cohort 3: Non-diseased Comparison Cohort
* Diagnosed for any serious chronic disease that is thought to adversely impact pregnancy.
* Exposed to a known human teratogen during pregnancy as confirmed by the OTIS Research Center

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women enrolled in the study will participate for the duration of that pregnancy. Those who deliver at least one live born infant and the infants will participate for 1 year after delivery of that infant.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Rate of major structural birth defect | Up to 1 year of age of the infant
  A major structural birth defect is a defect that has either cosmetic or functional significance to the child (eg, a cleft lip) and is identified up to one year of age by the mother, the health care provider/medical record, or identified in the dysmorphological examination.

SECONDARY OUTCOMES:
Pregnancy Outcomes: Spontaneous abortion | Date of conception to 20 weeks gestation
  Spontaneous abortion is defined as non-deliberate embryonic or fetal death that occurs < 20.0 weeks' gestation post-LMP (Last Menstrual period).
Pregnancy Outcomes: Stillbirth | After 20 weeks of gestation but prior to delivery
  Stillbirth is defined as a non-deliberate fetal death that occurs at or after 20 weeks of gestation but prior to delivery.
Pregnancy Outcomes: Premature delivery | Live birth prior to 37 weeks gestation
  Premature delivery is defined as live birth prior to 37 weeks' gestation as counted from LMP (Last Menstrual period).
Infant Outcomes: pattern of minor structural birth defects | Up to 1 year of age of the infant
  A specific pattern of 3 or more structural defects in live born infants with dysmorphological physical examination.
Infant Outcomes: Small for gestational age | At birth
  Proportion of infants less than or equal to the 10th percentile for sex and gestational age on weight, length, or head circumference.
Infant Outcomes: Postnatal growth deficiency | Up to 1 year of age of the infant
  Proportion of infants less than or equal to the 10th percentile for sex and age on weight, length, or head circumference at 1 year postnatal evaluation.
Infant Outcomes: Serious or opportunistic infections | Up to 1 year of age of the infant
  Proportion of infants who experienced serious or opportunistic infections up to 1 year of age.
Infant Outcomes: Hospitalizations | Up to 1 year of age of the infant
  Proportion of infants who experienced hospitalizations in the first year of life excluding those that are linked to premature delivery or birth defects included as endpoints.
Infant Outcomes: Malignancies | Up to 1 year of age of the infant -
  Proportion of infants who reported malignancies reported in an infant after birth and up to 1 year of age.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- United States, New York, New York, United States
- CANADA, Canada, Canada

IPD SHARING:
Plan to Share IPD: No